CLINICAL TRIAL: NCT01363635
Title: Severe Sepsis/Septic Shock on Admission to the General Surgical ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suneerat Kongsayreepong, MD, Professor, Mahidol University
Other Study IDs: Si199/2011
Record Dates: First submitted 2011-05-28; First posted 2011-06-01 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Septic Shock; Multiple Organ Failure; Fatal Outcome
Keywords: severe sepsis/septic shock; organ failure; AKI; PMI; ALI; Stroke; ICU death
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure; Sepsis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe sepsis: severe sepsis/septic shock, organ failure, ICU death

SUMMARY:
Severe sepsis/septic shock are serious complications of infection with high morbidity and mortality. Recent information showed that early and aggressive resuscitation may help improving survival and outcome especially the resuscitation within the first 3 hours. In surgical patients, either severe sepsis/septic shock bought them to the operating room or this sepsis might be found after surgery resulting in higher morbidity and mortality. Not only knowledge management, others possible risk factors should also be identified and corrected for outcome improving. This prospective observational study will be done in 800 adult surgical patients admitting to the general surgical intensive care unit. Incidence of severe sepsis/septic shock on admission along with risk factors associated with poor outcomes [organ failure (AKI, ALI, PMI, liver failure, stroke), prolonged ICU length of, stay, ICU death] will be recorded especially effect of amount and type of fluid replacement in the first 6 hours, 24, 48 and 72 hours after diagnosis. Outcome as major organ failure, ICU length of stay, ICU, 28 and 90 days mortality will also be study.

DETAILED DESCRIPTION:
Consecutive severe sepsis/ septic shock patients who will be admitted to the general surgical ICU of Siriraj Hospital, Mahidol University, Bangkok, Thailand will be recruited to this study. Apart from demographic data (age, sex, BMI, comorbidity), detail of septic shock and resuscitation (preoperative and intraoperative resuscitation), vasopressor and steroid used, type and amount of fluid, blood and blood component used and shock reversal time. Complication associated with surgery, anesthesia and in ICU will also recorded. Clinical outcome as organ failure (Stroke, PMI, aki, ARDS); ventilator day, ICU and hospital length of stay, mortality (in ICU, 28 and 90 days mortality) and cause of mortality will be carefully recorded

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years) surgical patient admitting to the general surgical ICU
* Consent to this study

Exclusion Criteria:

* Patient undergoing cardiothoracic surgery, neurosurgery and traumatic surgery
* Not consent to this study

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult surgical patient admiitiing to the general surgical ICU
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
incidence of severe sepsis/septic shock on admission to the general surgical ICU | 5 year
  Incidence of severe sepsis and septic shock on admission to the general surgical ICU

SECONDARY OUTCOMES:
risk factors associated with poor outcome (organ failure, prolonged ICU length of stay and ICU death) | 5 year
  organ failure (Stroke, AKI, PMI,ARDS), Mortality (ICU, 28 and 90 days) mortality and cause of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Suneerat Kongsayreepong, MD, Principal Investigator — Siriraj Hospital, Mahidol University, Bnagkok, Thailand
Locations (1):
- ICU Siamitra and ICU salad-Sumang, Deaprtment of Anesthesiology, Siriraj Hospital, Faculty of Medicine, Mahidol UNiversity, Bangkok, Thailand, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Result] Zahar JR, Timsit JF, Garrouste-Orgeas M, Francais A, Vesin A, Descorps-Declere A, Dubois Y, Souweine B, Haouache H, Goldgran-Toledano D, Allaouchiche B, Azoulay E, Adrie C. Outcomes in severe sepsis and patients with septic shock: pathogen species and infection sites are not associated with mortality. Crit Care Med. 2011 Aug;39(8):1886-95. doi: 10.1097/CCM.0b013e31821b827c. PMID 21516036